CLINICAL TRIAL: NCT00297817
Title: A Phase 2, Single-Blind, Controlled, Randomized Study of the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine ± OMV When Administered at an 0-2-6-Month Schedule in Healthy Adolescents 11-18 Years of Age
Brief Title: Study of the Safety and Immune Response of Two Serogroup B Meningococcal Vaccines Administered to Healthy Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V72P3
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-01

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal Disease; Meningococcal Meningitis; Vaccine
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: rMenB (Experimental)
  Interventions: Biological: serogroup B meningococcal vaccine
- Arm 2: rMenB + OMV (Experimental)
  Interventions: Biological: serogroup B meningococcal vaccine
- Arm 3: Placebo (Placebo Comparator)
  Interventions: Biological: serogroup B meningococcal vaccine

INTERVENTIONS:
Biological: serogroup B meningococcal vaccine — 0.5mL doses in pre-filled syringes. All subjects will receive the study vaccine following a 0,2,6 vaccination schedule.
  Arms: Arm 1: rMenB
Biological: serogroup B meningococcal vaccine — 0.5mL doses in pre-filled syringes. All subjects will receive the study vaccine following a 0,2,6 vaccination schedule.
  Arms: Arm 2: rMenB + OMV
Biological: serogroup B meningococcal vaccine — 0.5mL doses in pre-filled syringes. All subjects will receive the placebo following a 0,2,6 vaccination schedule.
  Arms: Arm 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of two serogroup B meningococcal vaccines in comparison to placebo administered to healthy adolescents ages 11 to 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adolescents between and including 11-18 years of age, who provide written informed consent.

Exclusion Criteria:

* Previous or suspected disease caused by N. meningitidis; or previous immunization with a serogroup B meningococcal vaccine; Any acute, chronic or progressive disease.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 2006-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and immunogenicity as measured by serum bactericidal activity of the two vaccines in healthy adolescents | 1 month after completion of immunization schedule

SECONDARY OUTCOMES:
Safety, tolerability and immunogenicity as measured by serum bactericidal activity of the two vaccines in healthy adolescents | 6 months after completion of immunization schedule

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Chair — Novartis
Locations (8):
- United States (8):
  - Encinitas, California
  - Atlanta, Georgia
  - St Louis, Missouri
  - Cleveland, Ohio
  - Galveston, Texas
  - Layton, Utah
  - Salt Lake City, Utah
  - Seattle, Washington